CLINICAL TRIAL: NCT05366335
Title: Value of Colonoscopic Probiotics Infusion in Patients With Functional Gastrointestinal Disease: a Prospective Randomized Controlled Study
Brief Title: Colonoscopic Probiotics Infusion for Functional Gastrointestinal Disease
Acronym: CPIFGD
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: First Affiliated Hospital Xi'an Jiaotong University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: XJTU1AF2022LSK-205
Record Dates: First submitted 2022-04-24; First posted 2022-05-09 (Actual); Last update posted 2022-08-04 (Actual); Status verified 2022-04

CONDITIONS: Functional Constipation; Irritable Bowel Syndrome; Probiotics; Colonoscopy
MeSH Terms: conditions — Irritable Bowel Syndrome | interventions — Lacteol; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Live Combined Bifidobacterium and Lactobacillus (Experimental): The experimental group receive basic treatment and a single infusion of Live Combined Bifidobacterium and Lactobacillus solution through colonoscopy.
  Interventions: Drug: Live Combined Bifidobacterium and Lactobacillus; Drug: Basic treatment
- Control (Placebo Comparator): The control group receive basic treatment and a single injection of normal saline through colonoscopy.
  Interventions: Drug: Normal saline; Drug: Basic treatment

INTERVENTIONS:
Drug: Live Combined Bifidobacterium and Lactobacillus — The invesitigators give patients Live Combined Bifidobacterium and Lactobacillus solution infusion during their colonoscopy examination for a single time in the Live Combined Bifidobacterium and Lactobacillus group.
  Other Names: Live combined Bifidobacterium and Lactobacillus solution infusion through colonoscopy
  Arms: Live Combined Bifidobacterium and Lactobacillus
Drug: Normal saline — The invesitigators give patients normal saline as a placebo infusion during their colonoscopy examination for a single time in the control group.
  Other Names: Normal saline as placebo infusion through colonoscopy
  Arms: Control
Drug: Basic treatment — The invesitigators give patients general treatment and drug treatment including oral Live Combined Bifidobacterium and Lactobacillus tablets as basic treatment.

SUMMARY:
The purpose of this project is to study the the efficacy and safety of probiotics implantation through infusion during colonoscopy in the treatment of functional constipation and irritable bowel syndrome. The study is a single-center, prospective, randomized, single-blind, controlled, cohort study. The invesitigators plan to enroll 80 patients with functional constipation and 80 patients with irritable bowel syndrome. The invesitigators will randomize the included study subjects. The experimental group receive basic treatment and a single infusion of probiotics through colonoscopy. The control group receive basic treatment and a single injection of normal saline through colonoscopy. The invesitigators will follow up the patients for 8-12 weeks. The primary endpoint is the efficacy of the single colonoscopic probiotics infusion in functional constipation and irritable bowel syndrome patients. The secondary endpoint is the safety of the single colonoscopic probiotics infusion in functional constipation and irritable bowel syndrome patients. Other exploratory objectives include the alterations in clinical indicators, fecal microbiota, and intestinal microbiota metabolites in feces and serum.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing for colonoscopy
* Meet Rome IV diagnostic criteria for functional constipation or irritable bowel syndrome
* Voluntarily participate in this clinical study and sign the informed consent.

Exclusion Criteria:

* Use of probiotics or antibiotics within the past 4 weeks
* History of intestinal surgery
* History of severe liver and kidney disease
* History of cardiovascular and cerebrovascular diseases
* History of neuropsychiatric diseases
* Pregnant women or lactating women
* Allergic to any ingredients of the live bacteria tablet

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2022-07-04 (Actual); Primary Completion 2022-10-31 (Estimated); Study Completion 2023-01-01 (Estimated)

PRIMARY OUTCOMES:
Proportion of effective patients with functional constipation and irritable bowel syndrome patients | 8-12 weeks after start of treatment.
  The efficacy of irritable bowel syndrome is evaluated by stool texture and abdominal discomfort related scales including IBS-SSS, BSS score, IBS-QOL,HADS and number of bowel movements per day in 12 weeks after start of treatment. The efficacy of functional constipation is evaluated by weekly defecation frequency, spontaneous complete bowel movement, and scales such as Wexner constipation score, BSS score, and PAC-QOL in 8 weeks after start of treatment.

SECONDARY OUTCOMES:
Incidence of adverse events related to treatment | 8-12 weeks after start of treatment.
  The safety of single colonoscopic probiotics infusion was evaluated by incidence of adverse events related to colonoscopic probiotics infusion during the treatment and 8-12 weeks after the treatment.

OTHER OUTCOMES:
Fecal microbiota | 8-12 weeks after start of treatment.
  16S rRNA detection of fecal intestinal flora.
Intestinal microbiota metabolites | 8-12 weeks after start of treatment.
  Detection of gut microbiota metabolites in blood and feces by HPLC-MS/MS.

CONTACTS AND LOCATIONS:
Overall Officials: Yun Feng, M.D., Study Chair — First Affiliated Hospital Xi'an Jiaotong University
Locations (1):
- First Affiliated Hospital of Xi'an Jiaotong University, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: No